CLINICAL TRIAL: NCT03203980
Title: Bleeding Events After Triple Antithrombotic Therapy Initiation: a Prospective Observational Study in Real Life
Brief Title: Bleeding Events After Triple Antithrombotic Therapy Initiation.
Acronym: HEMOTRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01733-50
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Triple antithrombotic therapy — patients who are prescribed double antiplatelets agents and oral anticoagulation (except VKA)

SUMMARY:
The optimal antithrombotic therapy for patients requiring anticoagulation after coronary stenting is unknown. Double platelets suppressive agents combined with oral anticoagulation (triple antithrombotic therapy) remains the Gold standard.

Our study aims at studying bleeding events occurring until 6 months after the initiation of triple antithrombotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring triple antithrombotic therapy, including double antiplatelets agents and oral anticoagulation

Exclusion Criteria:

* history of bleeding
* patients already under triple antithrombotic therapy
* patients under vitamin K antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the cardiology care unit of Nancy Central Hospital, hospitalised for coronary stenting and requiring oral anticoagulation (except VKA)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-07-15 (Estimated)

PRIMARY OUTCOMES:
Bleeding events | within 6 months since the initiation of triple antithrombotic therapy
  Bleeding events with clinical significance

IPD SHARING:
Plan to Share IPD: No